CLINICAL TRIAL: NCT05442632
Title: Director, Department of Liver Surgery, Fudan University Shanghai Cancer Center
Brief Title: Efficacy and Safety of Herombopag in Patients With Thrombocytopenia Before Hepatectomy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Lu Wang, MD, PhD, Chief physician, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OBU-SH-HCC-II-010
Record Dates: First submitted 2022-06-27; First posted 2022-07-05 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Hepatopathy
Keywords: Hepatopathy; thrombocytopenia; Hetrombopag
MeSH Terms: conditions — Digestive System Diseases; Thrombocytopenia | interventions — hetrombopag

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: 1 (Experimental): durg：Hetrombopag 5mg，once daily，oral
  Interventions: Drug: Hetrombopag
- Experimental: 2 (Experimental): Ndurg： Placebo 5mg，once daily，oral
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hetrombopag — The patients received Hetrombopag 5mg orally d1-14 days, surgery will be conducted at d6-14 day
  Arms: Experimental: 1
Drug: Placebo — The patients received Placebo 5mg orally d1-14 days, surgery will be conducted at d6-14 day
  Arms: Experimental: 2

SUMMARY:
This is a single center, randomized, controlled study, to evaluate the efficacy and safety of Herombopag in patients with Thrombocytopenia before hepatectomy.

DETAILED DESCRIPTION:
The purpose of this study is to assess the ability of Herombopag to elevate platelet counts thereby reducing the need for platelet transfusions in patients with thrombocytopenia before hepatectomy. The clinical benefit of Herombopag will be measured by the proportion of subjects who avoid platelet transfusions, before, during and up to 7 days after undergoing an hepatectomy. In addition, bleeding events will be monitored during this time. The number of transfusions, safety events will be monitored during this time and for up to 3 months after undergoing a hepatectomy to help further evaluate clinical benefit.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male and female subjects ≥18 years of age；
* 2.Patients prepared to receive hepatectomy；
* 3.50×10^9/L≤platelet count≤80×10^9/L；
* 4.Child-PUgh score A or grade B (≤7 )；
* 5.Life expectancy ≥3 months；
* 6.Normal Bone marrow hematopoiesis and renal function;
* 7.Voluntary participation and written informed consent;

Exclusion Criteria:

* 1.Central nervous system diseases caused by liver disease;
* 2.Platelet transfusion within 7 days prior to the first dose of study drug;
* 3.History of any primary hematologic disorder;
* 4.History of arterial or venous thrombosis, including thrombosis of any part of the splenic-mesenteric system;
* 5.Pre-diagnosed Immune Thrombocytopenic Purpura (ITP);
* 6.History of Myelodysplastic Syndrome (MDS);
* 7.Those with bleeding tendency，have evidence of hereditary bleeding or blood coagulation disorder;
* 8.Females who are pregnant (positive β-hCG test ) or breastfeeding;
* 9.Subjects who have participated in another investigational trial within 30 days prior to Visit 1;
* 10.Those with uncontrollable neurological and psychiatric diseases or mental disorders, poor compliance, unable to cooperate and describe treatment response;
* 11.Subjects with known intolerance or allergy to any of the ingredients in eltrombopag tablets;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2022-07-25 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients who require blood product infusion or intervention with platelet raising drugs due to bleeding during the perioperative period | From the start of using the investigational drug to 7 days after surgery completion
  Platelet transfusions were administered at the discretion of the investigator and the physician performing the hepatectomy.

SECONDARY OUTCOMES:
Proportion of patients with bleeding after surgery need intervention. | up to 7 days following surgery。
  The World Health Organization Bleeding Scale was used to assess bleeding following surgery.. The range of possible scores is 0 to 4. Grade 0 is no bleeding; Grade 1 is petechiae (small [1-2 millimeter] red or purple spot on the body, caused by a minor hemorrhage); Grade 2 is mild blood loss; Grade 3 is gross blood loss (requiring a transfusion; and Grade 4 is debilitating blood loss (retinal or cerebral associated with fatality).
Changes in preoperative Platelet count compared to baseline | baseline and up to 1 days prior to surgery
  Platelet count were determined from blood draws. platelet count collect on baseline and prior to 1 days of surgery. Missing platelet count assessments at any given time point was considered to be a non-response at that point and were not estimated
Proportion of patients whose Platelet count returned to ≥80×10^9/L | baseline and up to 1 days prior to surgery
  Platelet count were determined from blood draws. platelet count collect on baseline and prior to 1 days of surgery. Missing platelet count assessments at any given time point was considered to be a non-response at that point and were not estimated.
Incidence of deep venous thrombosis | up to 3 months following surgery.
  Imaging examination will be conducted at d1、d3、d5、d7、d14、end of one month、 end of three month after surgery, to evaluate deep venous thrombosis if necessary.
Incidence of liver failure | up to 3 months following surgery.
  Posthepatectomy liver failure is defined as: A postoperatively acquired deterioration in the ability of the liver to maintain its synthetic, excretory, and detoxifying functions, characterized by an increased international normalized ratio A postoperatively acquired deterioration in the ability of the liver to maintain its synthetic, excretory, and detoxifying functions, characterized by an increased international normalized ratio and hyperbilirubinemia on or after postoperative day 5. If international normalized ratio or serum bilirubin concentration is increased preoperatively, Post hepatectomy liver failure is defined by an increasing international normalized ratio and increasing serum bilirubin concentration on or after postoperative day 5 Other obvious causes for the observed biochemical and clinical alterations such as biliary obstruction should be ruled out. The evaluate of liver failure was conducted at d1、d3、d5、d7、d14、end of one month、 end of three month after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Lu Wang, Professor, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No